CLINICAL TRIAL: NCT05024357
Title: A Randomized Controlled Study of Tyrosine Kinase Inhibitor Maintenance Therapy Following Allogeneic Hematopoietic Stem Cell Transplantation in Newly Diagnosed Philadelphia Chromesome Positive Adult Acute Lymphoblastic Leukemia
Brief Title: A Study of TKI Maintenance Therapy Following Allo-HSCT in Newly Diagnosed Ph+ Adult ALL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2020-002-1
Record Dates: First submitted 2021-08-17; First posted 2021-08-27 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-08

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma; Philadelphia-Positive Acute Lymphoblastic Leukemia; ALL, Adult
Keywords: Philadelphia-Positive; Adult Acute Lymphoblastic Leukemia; Allogeneic Hematopoietic Stem Cell Transplantation; Tyrosine Kinase Inhibitors
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dasatinib for 1 year (Experimental): After the allo-HSCT treatment, the patients in this group will continue to take dasatinib orally for 1 year.
  Interventions: Drug: Dasatinib
- Dasatinib for 6 months (Experimental): After the allo-HSCT treatment, the patients in this group will receive dasatinib for 6 months.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Take Dasatinib orally for 1 year or 6 months post-HSCT.
  Other Names: Dasatinib tablet

SUMMARY:
This project is a key clinical research project approved by the Clinical Research Center of the First Affiliated Hospital of Xi 'an Jiaotong University.Tyrosine kinase inhibitors (TKI) combined with chemotherapy and subsequent allogeneic hematopoietic stem cell transplantation (allo-HSCT) are routinely used in patients with philadelpha-positive lymphoblastic leukemia (Ph+ALL). However, TKI maintenance therapy post-HSCT remains controversial. In this study, Ph+ALL patients are enrolled and given dasatinib combined with chemotherapy followed by allo-HSCT. Then patients in the group A continuing to use dasatinib for 1 year is compared with those in the group B receiving dasatinib for 6 months after HSCT. The measurable residual disease (MRD), complete remission (CR), overall survival (OS), disease free survival (DFS), non-relapse mortality (NRM) and the incidence of graft versus host disease (GVHD) will be observed to determine the optimal duration of TKI maintenance therapy post-HSCT.

DETAILED DESCRIPTION:
About 25% of adult patients with acute lymphoblastic leukemia (ALL) are associated with t (9; 22), positive philadelphia chromosome (Ph+ ALL), in whom BCR/ABL fusion gene can be detected in the bone marrow and peripheral blood. Although current treatment strategies using tyrosine kinase inhibitors (TKIs) such as dasatinib combined with chemotherapy have achieved high complete remission (CR) rates, the duration of remission is short, and most Ph+ ALL patients relapse within 2 years. Allogeneic hematopoietic stem cell transplantation (allo-HSCT) bridging to CR remains the only strategy to cure Ph+ ALL. However, TKI maintenance therapy post-HSCT remains controversial. In this study, Ph+ALL patients are enrolled. The participants will receive dasatinib combined with induction and consolidation chemotherapy to obtain molecular remission and then undergo allo-HSCT. After the above treatments, the patients will be randomly divided into two groups. The subjects in the group A will continue to use dasatinib for 1 year, while the patients in the group B receive dasatinib for 6 months post-HSCT. The measurable residual disease (MRD), CR, overall survival (OS), disease free survival (DFS), non-relapse mortality (NRM) and the incidence of graft versus host disease (GVHD) will be observed to determine the optimal duration of TKI maintenance therapy post-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old, newly diagnosed as Ph+ALL.
* Sign the informed consent.
* Have appropriate allo-HSCT donors.
* Accept allo-HSCT.
* Accept follow-up.

Exclusion Criteria:

* Liver and kidney function impairment: serum transaminase > 2 times of the upper limit of normal value, total bilirubin > 1.5 times of the upper limit of normal value, serum inosine > the upper limit of normal value (97 umol/L).
* Active hepatitis B, hepatitis C or tuberculosis infection.
* Can not tolerate the adverse effects of dasatinib.
* Pregnancy.
* Diagnosis of mental disorders.
* Failed to reach molecular complete remission (MCR) after the early treatment.
* Do not accept follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients with Measurable Residual Disease (MRD) Positivity | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  MRD means the subclinical levels of residual leukemia.
Percentage of Patients with Complete Remission (CR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  CR means that the blood counts have returned to normal, the leukemia cannot be seen when a bone marrow sample is examined under the microscope, and the signs and symptoms of the ALL are gone.

SECONDARY OUTCOMES:
Disease-free Survival (DFS), months | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  The measure of time after allo-HSCT during which no sign of ALL is found.
Overall Survival (OS), months | From date of randomization until the date of death from any cause, whichever came first, assessed up to 36 months.
  The length of time from the date of allo-HSCT that Ph+ ALL patients are still alive.
Non-relapse Mortality (NRM), rate or percentage | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  NRM means death without recurrent or progressive disease after allo-HSCT.
Incidence of graft versus host disease (GVHD), rate or percentage | From date of randomization until the date of GVHD occurrence or date of death from any cause, whichever came first, assessed up to 36 months.
  GVHD is a condition that might occur after allo-HSCT. In GVHD, the donated bone marrow or peripheral blood stem cells view the recipient's body as foreign, and the donated cells/bone marrow attack the body.
Adverse Effects (AE) | From date of randomization until the date of death from any cause, whichever came first, assessed up to 36 months.
  An adverse effect is any untoward medical occurrence in clinical investigation subject administered dasatinib and which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pengcheng He, Study Chair — First Affiliated Hospital of Xian Jiaotong University; Xiaoning Wang, Study Director — First Affiliated Hospital of Xian Jiaotong University; Huachao Zhu, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University; Juan Ren, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University; Ying Chen, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University; Ting Fan, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China